CLINICAL TRIAL: NCT03299842
Title: An Exploratory, Pilot Study to Assess the Usability of the Embrace Seizure Detection Watch in Children and Young Adults With Dravet Syndrome: A Sub-study to the ZX008-1503 Open-Label Extension Trial
Brief Title: A Study to Assess the Usability of the Embrace Seizure Detection Watch in Children and Young Adults With Dravet Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to low enrollment.
Sponsor: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX008-1503-SS01
Record Dates: First submitted 2017-09-10; First posted 2017-10-03 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Dravet Syndrome
Keywords: seizure; tonic clonic; epilepsy; myoclonic; encephalopathy
MeSH Terms: conditions — Epilepsies, Myoclonic; Seizures; Epilepsy; Brain Diseases | interventions — Fenfluramine

STUDY DESIGN:
Intervention Model Description: ZX008-1503 Fenfluramine, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZX008 (Experimental): ZX008 is supplied as an oral solution in a concentration of 2.5 mg/mL. Subjects will be titrated to an effective dose beginning with 0.2 mg/kg/day (maximum: 30 mg/day).
  Interventions: Drug: ZX008 (Fenfluramine Hydrochloride)

INTERVENTIONS:
Drug: ZX008 (Fenfluramine Hydrochloride) — ZX008 is supplied as an oral solution in a concentration of 2.5 mg/mL. Subjects will be titrated to an effective dose beginning with 0.2 mg/kg/day (maximum: 30 mg/day).

SUMMARY:
This is an exploratory sub-study to ZX008-1503 [NCT02823145]. Subjects will be fitted with an Embrace seizure detection watch and seizures detected by the watch will be compared to those entered into an electronic seizure diary.

DETAILED DESCRIPTION:
This sub study will include up to 20 participants who meet the entry criteria for the main Study ZX008-1503 and who are willing to wear the Embrace watch and use the Embrace Alert app for 12 consecutive weeks. Those invited to participate will undergo all procedures included in the main study during their participation in this sub-study,

ELIGIBILITY:
Inclusion Criteria:

* Meeting all of the main study ZX008-1503 [NCT02823145] inclusion criteria
* Subject is willing to wear the Embrace watch on the wrist (alternatively ankle, if needed for younger children). Subjects are asked to wear the watch for as many hours of the day as possible and for the entire night, if possible, for the duration of the sub-study.
* Subject's parent/caregiver is willing to use the Alert App.
* Subject/subject's caregiver is willing to ensure that the Embrace watch remains within close proximity of the paired iPod Touch running the Empatica Alert app.

Exclusion Criteria:

* Subject has a known hypersensitivity to any of the Embrace device materials.
* Subject has a clinically significant condition, or has had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to Visit 1, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the subject.

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - The Children's Hospital Colorado, Aurora, Colorado

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This exploratory sub-study started to enroll participants in July 2017 and concluded in July 2018. Investigating a rare disease in pediatrics, this exploratory sub-study was terminated due to low enrolment. Of the 20 participants the Sponsor attempted to enroll in the study, only 5 participants enrolled and terminated early from the study.
Groups:
- ZX008: Participants received ZX008 (fenfluramine hydrochloride) as an oral solution in a concentration of 2.5 milligrams per milliliter (mg/mL). Participants were titrated to an effective dose beginning with 0.2 milligrams per kilogram per day (mg/kg/day) to maximum dose of 30 mg/day. Study medication was administered twice a day (BID) in equally divided doses with food for 12 consecutive weeks, as per main study protocol, ZX008-1503 [NCT02823145]. For this substudy, ZX008-1503-SS01, all participants were required to wear the noninvasive Empatica Embrace watch system (EMBRACE) wrist-worn monitoring device.
Period: Overall Study
Arm/Group | ZX008
Started | 5
Completed | 0
Not Completed | 5
Not completed — Caregiver withdrew consent | 2
Not completed — Child would not keep the watch on | 3

BASELINE CHARACTERISTICS:
Population: No data will be reported, as the study was investigating a rare disease in pediatrics with a high risk of participant identification due to low enrolment (participant privacy/confidentiality issue).
Arm/Group | ZX008
Number analyzed (Participants) | 0
Age, Categorical [unit: participants]
Age, Continuous [unit: years]
Sex: Female, Male [unit: participants]
Race/Ethnicity, Customized [unit: participants]
Race/Ethnicity, Customized [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Overall Usability of the Empatica Embrace Seizure Detection Watch System (Embrace) in Outpatients With Dravet Syndrome
Description: The assessment of user experience with Embrace watch system included Likert Ease of Use Questionnaire. The questionnaire had 3 items related to use of the Embrace watch, Mate App and Alert App. All the questions were responded on 5-point Likert scale (1-Very difficult, 2-difficult, 3-Neutral, 4-Easy and 5-Very easy). Response to each item on the questionnaire was reported. Responses across all items on the questionnaire were summed to create an overall index with total score of 0 to 15, where higher scores represents the better usability of the device.
Time Frame: Approximately 12 weeks
Population: as for baseline characteristics
Arm/Group | ZX008
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 12 weeks
Description: No data will be reported, as the study was investigating a rare disease in pediatrics with a high risk of participant identification due to low enrolment (participant privacy/confidentiality issue).
Arm/Group | ZX008
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No data will be reported, as the exploratory sub-study was investigating a rare disease in pediatrics with a high risk of participant identification due to low enrolment (participant privacy/confidentiality issue). Safety Data for eligible participants in the sub-study was collected in the main study ZX008-1503 (NCT02823145) as pre-specified in the protocol. The data will be disclosed with the main study results posting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT03299842/Prot_SAP_003.pdf